CLINICAL TRIAL: NCT05680623
Title: Clinical and Economic Validation of the International Study Group for Pancreatic Surgery (ISGPS) Definition of Postpancreatectomy Acute Pancreatitis (PPAP)
Brief Title: Clinical and Economic Validation of the ISGPS Definition of PPAP
Acronym: ISGPS-PPAP
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Collaborators: Heidelberg University (Other); Catholic University of the Sacred Heart (Other); Hospices Civils de Lyon (Other); Lund University (Other); Flinders Medical Centre (Other Government); Amsterdam UMC, location VUmc (Other); University of Dublin, Trinity College (Other); Christchurch Hospital (Other); University of Colorado, Denver (Other); Scientific Institute San Raffaele (Other); University of Graz (Other); Technical University of Munich (Other); Royal Free Hospital NHS Foundation Trust (Other); San Gerardo Hospital (Other); University of Liverpool (Other); Universitätsklinikum Hamburg-Eppendorf (Other); Massachusetts General Hospital (Other); Kyushu University (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Petz Aladar County Teaching Hospital (Other); Mayo Clinic (Other); Hospital Miguel Servet (Other); Tata Memorial Hospital (Other Government); Medical University of Vienna (Other); Kyoto University, Graduate School of Medicine (Other); UnitedHealth Group (Industry); Ludwig-Maximilians - University of Munich (Other); Thomas Jefferson University (Other); Humanitas Hospital, Italy (Other); Indiana University Health (Other); University of Manchester (Other); New York University (Other)
Responsible Party: Sponsor
Other Study IDs: 3822CESC
Record Dates: First submitted 2022-10-19; First posted 2023-01-11 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Postoperative Acute Pancreatitis; Pancreaticoduodenectomy; Postoperative Pancreatic Fistula; Postoperative Complications
Keywords: pancreatitis; hyperamylasemia; pancreatoduodenectomy; postoperative complications; pancreatic fistula
MeSH Terms: conditions — Postoperative Complications; Pancreatitis; Hyperamylasemia; Pancreatic Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study population: Subgroups based on the ISGPS diagnostic criteria and the grading system of PPAP:
  1. Without PPAP or POH: Patients without POH nor imaging consistent with AP.
  2. POH: sustained postoperative serum hyperamylasemia neither clinically relevant nor consistent imaging
  3. PPAP: requiring the fulfilment of three criteria:
     * POH: sustained serum hyperamylasemia greater than the institutional upper limit of normal persisting on postoperative days 1 and 2;
     * macroscopic radiologic features of AP
     * clinically relevant complications. PPAP severity will be classified into grades B and C, with progressive clinical deterioration.
  Interventions: Diagnostic Test: PPAP diagnosis

INTERVENTIONS:
Diagnostic Test: PPAP diagnosis — Serum amylase (total or the pancreatic isoform) and/or lipase activity will be systematically measured at least on postoperative days 1 and 2.
  A CT with pancreas protocol iv contrast infusion will be performed in the postoperative course when clinically required, facing patients' clinical worsening, suspicious of abdominal complications.

SUMMARY:
This prospective validation study aims to investigate the incidence of PPAP after pancreaticoduodenectomy (PD) by applying the ISGPS definition and grading system, to demonstrate its clinical impact by examining associated postoperative outcomes, and to validate its applicability through an economic assessment.

DETAILED DESCRIPTION:
The study will be conducted at approximately 37 investigative sites in Europe, Asia, Oceania, and the United States. Only high volume centers for Pancreatic Surgery will be included in the study. All patients scheduled to receive elective pancreaticoduodenectomy (PD Kausch-Whipple or Longmire-Traverso) for all type of pancreatic disease (benign, malignant, or premalignant) will be enrolled. The study duration per subject will be up to 30 days after surgery or all the in-hospital lengths of stay. Preoperative care will follow institutional standards, according to each center involved. Surgical resection and reconstruction will be carried out according to the techniques adopted by each participating center. Both patients undergoing open and minimally invasive surgery can be considered eligible. Postoperative management will follow the institutional standards of each center. Serum amylase (total or the pancreatic isoform) and/or lipase activity will be systematically measured at least on postoperative days (POD) 1 and 2.Serum C-reactive protein (CRP) will be measured according to each institutional policy and reported once assessed from POD 1 to 3. Drain fluid amylase, or lipase activity will be checked according to the Institutional standards of each involved, and the values will be retrieved whether assessed from POD 1 to five. Radiological imaging will be performed in the postoperative course when clinically required, facing patients' clinical worsening, suspicious for abdominal complications.The severity of complications will be assessed according to the Clavien-Dindo (CD) classification system 32 . Readmission will be defined as a new hospital admission after discharge within 30 days from index surgery. Length of hospital stay is calculated from the day of surgery to discharge. Preoperative, intra-operative, and postoperative data will be recorded prospectively.

The estimated study duration will be 15 months. Time for data analysis must be considered negligible. Patients' follow-up will last 30 days after surgery to catch any additional morbidity even after discharge from the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective PD;
* Male and females ≥ 18 years;
* Upfront or after neoadjuvant therapy surgery is allowed;
* The ability of the subject to understand the character and individual consequences of the clinical trial;
* Written informed consent.

Exclusion Criteria:

* Patients undergoing emergency surgery;
* Informed consent withdrawal;
* Inability to perform the resection for any reason;
* Total or distal pancreatectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients scheduled to receive elective pancreaticoduodenectomy (PD - Kausch-Whipple or Longmire-Traverso) for all type of pancreatic disease (benign, malignant, or premalignant) will be enrolled.
Sampling Method: Probability Sample
Enrollment: 2900 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-01-12 (Actual)

PRIMARY OUTCOMES:
The incidence of PPAP | 30 postoperative days
  The incidence of PPAP after pancreaticoduodenectomy (PD) by applying the ISGPS definition and grading system.
The incidence of unplanned ICU admissions and hospital readmission in the PPAP group compared to the non-PPAP one. | 30 postoperative days
  Only an unplanned need for intensive care will be defined as intensive care unit (ICU) stay. Readmission will be defined as a new hospital admission after discharge within 30 days from index surgery.
The difference in length of hospital stay between the PPAP and the non-PPAP group | up to hospital discharge, an average of 30 postoperative days
  Length of hospital stay is calculated from the day of surgery to discharge.
The difference in hospital costs among the different grades of severity according to the ISGPS grading system22: no PPAP or POH, POH, PPAP grade B, and PPAP grade C groups. | 30 postoperative days
  Total hospital costs will comprise the cost of the index admission and every surgery-related readmission within 30 days from the index surgery. Costs will be inflation-adjusted using the standardized national consumer price index and normalized to adjust the variability inherent to different health systems and institutions.

SECONDARY OUTCOMES:
Correlation between postoperative serum amylase/serum lipase activity (U/L) and radiologic feature consistent with PPAP retrieved at postoperative imaging. | 30 postoperative days
  Serum amylase and/or lipase activity will be systematically measured on postoperative days (POD) 1 and 2.
  Radiological imaging will be performed in the postoperative course when clinically required, facing the patient's clinical worsening, and suspicious of abdominal complications.
Incidence and descriptive analysis of radiological features consistent with PAPP at postoperative imaging retrieved at different time points. | 30 postoperative days
  The radiologic evaluation will include the pancreas enlargement, pancreas enhancement, pancreatic necrosis and percentage, peripancreatic collections, characteristics, and their location, haemorrhage and pseudoaneurysm, ascites, thrombosis, main pancreatic duct diameter (mm), POD imaging (days).
Incidence and severity of postoperative morbidity. | 30 postoperative days
  Postoperative morbidity will be defined according to ISGPS definitions of postoperative pancreatic fistula, delayed gastric emptying, post-pancreatectomy hemorrhage, and chyle leak. Bile leakage as defined by ISGLS. Acute kidney injury will be determined according to 2012 Kidney Disease: Improving Global Outcomes (KDIGO) guidelines. The severity of complications will be assessed according to the Clavien-Dindo classification system.
Incidence of postoperative mortality. | 30 postoperative days
  Mortality will be defined as postoperative death recorded out to the point of 30-days postoperatively. Beyond these time limits, the mortality, possibly related to PPAP, will be considered and discussed in each case.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Marchegiani, Principal Investigator — Azienda Ospedaliera Universitaria Integrata di Verona
Locations (1):
- Giovanni Marchegiani, Verona, Italy

REFERENCES:
- [Background] Marchegiani G, Barreto SG, Bannone E, Sarr M, Vollmer CM, Connor S, Falconi M, Besselink MG, Salvia R, Wolfgang CL, Zyromski NJ, Yeo CJ, Adham M, Siriwardena AK, Takaori K, Hilal MA, Loos M, Probst P, Hackert T, Strobel O, Busch ORC, Lillemoe KD, Miao Y, Halloran CM, Werner J, Friess H, Izbicki JR, Bockhorn M, Vashist YK, Conlon K, Passas I, Gianotti L, Del Chiaro M, Schulick RD, Montorsi M, Olah A, Fusai GK, Serrablo A, Zerbi A, Fingerhut A, Andersson R, Padbury R, Dervenis C, Neoptolemos JP, Bassi C, Buchler MW, Shrikhande SV; International Study Group for Pancreatic Surgery. Postpancreatectomy Acute Pancreatitis (PPAP): Definition and Grading From the International Study Group for Pancreatic Surgery (ISGPS). Ann Surg. 2022 Apr 1;275(4):663-672. doi: 10.1097/SLA.0000000000005226. PMID 34596077
- [Background] Bannone E, Andrianello S, Marchegiani G, Masini G, Malleo G, Bassi C, Salvia R. Postoperative Acute Pancreatitis Following Pancreaticoduodenectomy: A Determinant of Fistula Potentially Driven by the Intraoperative Fluid Management. Ann Surg. 2018 Nov;268(5):815-822. doi: 10.1097/SLA.0000000000002900. PMID 30004917
- [Background] Loos M, Strobel O, Dietrich M, Mehrabi A, Ramouz A, Al-Saeedi M, Muller-Stich BP, Diener MK, Schneider M, Berchtold C, Feisst M, Hinz U, Mayer P, Giannakis A, Schneider D, Weigand MA, Buchler MW, Hackert T. Hyperamylasemia and acute pancreatitis after pancreatoduodenectomy: Two different entities. Surgery. 2021 Feb;169(2):369-376. doi: 10.1016/j.surg.2020.07.050. Epub 2020 Sep 25. PMID 32981689
- [Background] Chen H, Wang W, Ying X, Deng X, Peng C, Cheng D, Shen B. Predictive factors for postoperative pancreatitis after pancreaticoduodenectomy: A single-center retrospective analysis of 1465 patients. Pancreatology. 2020 Mar;20(2):211-216. doi: 10.1016/j.pan.2019.11.014. Epub 2019 Nov 27. PMID 31831390
- [Background] Partelli S, Tamburrino D, Andreasi V, Mazzocato S, Crippa S, Perretti E, Belfiori G, Marmorale C, Balzano G, Falconi M. Implications of increased serum amylase after pancreaticoduodenectomy: toward a better definition of clinically relevant postoperative acute pancreatitis. HPB (Oxford). 2020 Nov;22(11):1645-1653. doi: 10.1016/j.hpb.2020.03.010. Epub 2020 Apr 11. PMID 32291175